CLINICAL TRIAL: NCT04725344
Title: Relevance of the Activ'Dos App for Chronic Low Back Pain Patients - Randomized Trial
Brief Title: Relevance of the Activ'Dos App for Chronic Low Back Pain Patients
Acronym: ACTIV'DOS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitement difficulties
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 29BRC20.0294
Record Dates: First submitted 2021-01-04; First posted 2021-01-26 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: Chronic Disease; Lumbago
Keywords: Exercise; Self-rehabilitation; Chronic low back pain; Mobile app; mHealth; eHealth; Physiotherapy; Disability; Pain
MeSH Terms: conditions — Chronic Disease; Low Back Pain; Motor Activity; Pain

STUDY DESIGN:
Intervention Model Description: There are 2 groups : an interventional group with ACTIV'DOS app ; and a control group with a standard procedure using a sheet of paper.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACTIV'DOS group (Experimental): ACTIV'DOS is a smartphone application of self rehabilitation. There are 7 muscular exercices. Patients going to exercices during 15 minutes per day, during 6 weeks.
  Interventions: Other: ACTIV'DOS group
- Control group (Experimental): This group uses a sheet of paper for self-rehabilitation exercise. The self-rehabilitation program is the same as the ACTIV'DOS group. Patients have to exercise during 15 minutes per day, during 6 weeks.
  Interventions: Other: Usual practise

INTERVENTIONS:
Other: ACTIV'DOS group — ACTIV'DOS group use ACTIV'DOS application (with smartphone) to do the self rehabilitation each day (15 minutes per day) during 6 weeks. There are 7 exercices.
  Arms: ACTIV'DOS group
Other: Usual practise — Control group uses a standard sheet of paper to do the self-rehabilitation (15 minutes per day) during 6 weeks. There are 7 exercises.
  Arms: Control group

SUMMARY:
The purpose of this study is to compare a self rehabilitation program using ACTIV'DOS app versus using a standard sheet of paper.

DETAILED DESCRIPTION:
This study involves patients with chronic low back pain. The purpose of this study is to compare a self-rehabilitation program using ACTIV'DOS app versus a standard sheet of paper. Disabilities are measured with a Roland-Morris questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* chronic low back pain for more than 3 months
* Aged to 18 or more
* Possibility to use Activ'dos application with smartphone or tablet
* Initial score of Roland Morris questionnaire >= 4
* Fit to consent
* Who has signed consent form

Exclusion Criteria:

* Any signs of severe illness underlying to radicular and lumbar pain like red flags
* Guardianship or protection of vulnerable adult
* Pregnant or nursing
* Refuse to participate

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-05-09 (Actual)

PRIMARY OUTCOMES:
Change from functional impairment with Roland-Morris questionnaire at 6 weeks. | Day 0 (patient inclusion) and Day 42 (end of patient monitoring)
  Disabilities are measured with Roland-Morris questionnaire, from Day 0 to Day 42. This questionnaire includes 24 items with 1 point per item. The score ranges from 0 (no disability) to 24 (max. disability).

SECONDARY OUTCOMES:
Difference of average pain during the seven last days with VAS pain | Day 0 (patient inclusion) and Day 42 (end of patient monitoring)
  VAS pain is a scale measuring pain intensity from 0 (no pain) to 10 (extreme pain). For this outcome, the average pain during the seven last days is evaluated.
Difference of worse pain during the seven last days with VAS pain | Day 0 (patient inclusion) and Day 42 (end of patient monitoring)
  VAS pain is a scale measuring pain intensity from 0 (no pain) to 10 (extreme pain). For this outcome, the worse pain during the seven last days is evaluated.
Compliance (number of sessions done over the number of recommanded sessions) of self-rehabilitation program at 6 weeks | Day 42 (end of patient monitoring)
  Compliance is evaluated with a compliance table. Patients have to complete this table after each session. Investigators will report the compliance table at the end of the patient monitoring (Week 6).
Assessment of satisfaction with Likert scale | Day 42 (end of patient monitoring)
  Likert scale is a scale with 10 questions. For each question, the scale ranges from 3 (strongly agree) to -3 (strongly disagree).

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Cabinet de kinésithérapie Natanaël AUDREN, Brest
  - Cabinet de kinésithérapie Pierre VAL, Brest
  - Cabinet de kinésithérapie Pol KEROUANTON, Brest
  - Cabinet de kinésithérapie Vincent LUCAS, Brest

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest University Hospital. Requestors will be required to sign and complete a data access agreement.